CLINICAL TRIAL: NCT01877785
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MHAA4549A in Healthy Volunteers
Brief Title: A Study of MHAA4549A to Assess Safety And Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GV28916
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gedivumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MHAA4549A Arm (Experimental)
  Interventions: Drug: MHAA4549A
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHAA4549A — Single-ascending dose of MHAA4549A
  Arms: MHAA4549A Arm
Drug: Placebo — Placebo to MHAA4549A
  Arms: Placebo Arm

SUMMARY:
This randomized, double-blind, placebo-controlled, single-ascending dose study will assess the safety, tolerability and pharmacokinetics of ascending doses of MHAA4549A in healthy volunteers. Volunteers will be randomized to receive a single dose of MHAA4549A or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive
* Weight 40 to 100 kg
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations should be within the reference range for the test laboratory unless deemed not clinically significant by the investigator and Sponsor
* Volunteers agree to use acceptable contraceptive measures

Exclusion Criteria:

* History or clinically significant manifestations of disorders
* History of anaphylaxis, hypersensitivity or drug allergies
* History or presence of an abnormal ECG
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit
* History of significant drug abuse within 1 year prior to screening
* Current tobacco smokers
* Positive drug screen at screening or at check-in
* Positive pregnancy test result at screening or Day -1 or breast feeding during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 120 days

SECONDARY OUTCOMES:
Incidence of anti-therapeutic antibodies | 120 days
Pharmacokinetics: Serum concentration-time profile of MHAA4549A | Pre-dose on day 1 to day 120 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Québec, Quebec, Canada

REFERENCES:
- [Derived] Lim JJ, Deng R, Derby MA, Larouche R, Horn P, Anderson M, Maia M, Carrier S, Pelletier I, Burgess T, Kulkarni P, Newton E, Tavel JA. Two Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Studies To Investigate the Safety, Tolerability, and Pharmacokinetics of an Anti-Influenza A Virus Monoclonal Antibody, MHAA4549A, in Healthy Volunteers. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5437-44. doi: 10.1128/AAC.00607-16. Print 2016 Sep. PMID 27381392